CLINICAL TRIAL: NCT04073316
Title: AntiCoagulants and COGnition (ACCOG Trial): a Single-blind Randomized Controlled Trial Comparing the Neurocognitive Effects of Rivaroxaban Versus Vitamin K Antagonist
Brief Title: AntiCoagulants and COGnition
Acronym: ACCOG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-000794-23
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Nonvalvular Atrial Fibrillation
MeSH Terms: interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Intervention" group (Experimental)
  Interventions: Drug: Rivaroxaban 20 MG
- "Control" group (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban 20 MG — Rivaroxaban intake, 20mg/day
  Arms: "Intervention" group
Drug: Warfarin — Warfarin intake, with target INR range between 2 and 3
  Arms: "Control" group

SUMMARY:
The purpose of this study is to compare the change of global cognitive performance after 52 weeks of intervention among participants with nonvalvular atrial fibrillation (NVAF) receiving rivaroxaban versus a vitamin K antagonist (warfarin).

The secondary objectives are to compare, among participants with NVFA receiving rivaroxaban versus warfarin :

* the changes of global cognitive performance after 26 weeks of intervention
* the changes of executive functions after 26 and 52 weeks of intervention
* the changes of episodic memory after 26 and 52 weeks of intervention
* the changes of independence and autonomy after 26 and 52 weeks of intervention

DETAILED DESCRIPTION:
Detailed Description:

Vitamin K antagonists (VKAs) are commonly used for their role in hemostasis by interfering with vitamin K cycle decreasing the bioavailability of the vitamin K active form. In addition to a role in blood coagulation, vitamin K participates in brain health and function by regulating the synthesis of sphingolipids, a constituent of the myelins sheath and the neurons membrane, and through the biological activation of vitamin K-dependent proteins (VKDPs) involved in neuron survival. Epidemiological studies have reported a positive association between higher serum vitamin K concentration and better verbal episodic memory performance in older adults, and an inverse association between dietary vitamin K intakes and behavioural disorders and cognitive complaint. The clinical implication is that the use of VKAs, which deplete the active form of vitamin K, may be responsible for Central Nervous System (CNS) disorders.

CNS abnormalities were observed in newborns exposed in utero to VKA. Similarly, the investigators and other researchers reported that the use of VKAs (especially fluindione) was directly associated with cognitive decline (notably executive dysfunction) and hippocampal atrophy in older adults, even while taking into account the history of atrial fibrillation, stroke and vascular brain changes. These cross-sectional and longitudinal studies were yet limited by their observational design. Clinical trials are now warranted to explore the effect on cognition of VKAs against direct oral anticoagulants (DOACs), whose indications are similar but whose mechanism does not interfere with vitamin K. The favorable impact of the use of DOACs compared to VKA in the incidence of dementia was also observed in a US retrospective population-based study of patients managed per routine clinical care.

The investigators hypothesize that VKAs have a deleterious impact on cognition and brain morphology compared to DOACs, due to the decrease in vitamin K bioavailability. A review of the published clinical trials comparing the effects of VKAs and DOACs, especially rivaroxaban, shows that cognition and brain volume were not assessed as outcomes in these trials.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 70 years old
* Newly diagnosed hemodynamically stable NVAF longer than 52 hours or of unknown duration, and CHA2DS2-VASc score according to ESC 2016 guidelines for anticoagulation treatment indications
* MMSE score ≥ 20
* Subjects who can give written consent to participate in the study
* Affiliation to a social security scheme.

Exclusion Criteria:

* Known history of stroke and/or a diagnosed condition of dementia (DSM-IV criteria) and/or severe depressive symptomatology (score on the 4-item Geriatric Depression Scale > 3)
* Moderate or severe mitral stenosis
* Conditions other than NVAF that require anticoagulation
* Use of anticoagulant more than 3 days at inclusion or more than 15 days in the preceding 12 months
* Regular use of antiplatelet medications and/or nonsteroidal anti-inflammatory agents and/or azole class of antifungal agents and/or inhibitor of HIV protease
* Acute thromboembolic events or thrombosis (venous/arterial) within the last 14 days prior to randomization
* Known presence of cardiac thombus or myxoma or valvular atrial fibrillation
* Any contraindication to anticoagulation, high risk of bleeding, and any other contraindication listed in the local labeling for the experimental treatment and comparator treatment
* Unstable health, severe hepatic failure, or severe and moderate renal failure (creatinine clearance <50 mL/min), acute coronary syndromes
* Participation in another simultaneous clinical trial
* Inability to understand and speak French
* Refusal to participate from the participant
* Persons deprived of their liberty by administrative or judicial decision, persons under psychiatric care under duress, adults subject to a legal protection measure or unable to express their consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive performance | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Global cognitive performance is assessed with Alzheimer's Disease Assessment Scale-cognition score (ADAS-cog).
  Total scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment.

SECONDARY OUTCOMES:
Change in executive functions | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Executive functions are assessed with Frontal Assessment Battery score (FAB).
Change in executive functions | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Executive functions are assessed with digit spans.
Change in executive functions | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Executive functions are assessed with Trail Making Tests (TMT) parts A and B.
Change in executive functions | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Executive functions are assessed with Stroop test.
Change in executive functions | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Executive functions are assessed with the Processing Speed Index.
Change in episodic memory | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Episodic memory is assessed with Five-word test. The 5-word test studies the recall of a short list. The score of the first immediate recall and the score of the delayed recall should normally be equal to 10.
Change in independence and autonomy | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Independence and autonomy are assessed with Activities of Daily Living (ADL) score.
  ADL is an autonomy assessment grid (from 0 to 6) for basic activities of daily living (ADL).
  The lower the score, the more dependent the patient is.
Change in independence and autonomy | This outcome is assessed at baseline, 26 and 52 weeks after inclusion.
  Independence and autonomy are assessed with the 4-item Instrumental Activities of Daily Living (IADL-PAQUID) score.
  This test is used to assess the level of dependence in instrumental activities of daily living.
  The scale ranges from 0 to 4, with 0 indicating total dysautonomy and 4 indicating a totally autonomous person.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France